CLINICAL TRIAL: NCT01781091
Title: S4 :RANDOMIZED CONTROLLED TRIAL OF FULLY CLOSED-LOOP VENTILATION IN ICU.
Brief Title: S4 :Trial Of Fully Closed-Loop Ventilation In ICU.
Acronym: S4
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CH-2012-02; 2012-A1069-34 (Other: ANSM( France))
Record Dates: First submitted 2013-01-24; First posted 2013-01-31 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Intensive Care Patients Invasively Ventilated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- FULLY CLOSED-LOOP VENTILATION (Experimental): IntelliVent-ASV automatic mode
  Interventions: Device: INTELLIVENT ASV FULLY CLOSED-LOOP VENTILATION
- Conventional modes ventilation (Active Comparator): Conventional modes
  Interventions: Device: Conventionals Modes

INTERVENTIONS:
Device: INTELLIVENT ASV FULLY CLOSED-LOOP VENTILATION
  Arms: FULLY CLOSED-LOOP VENTILATION
Device: Conventionals Modes
  Arms: Conventional modes ventilation

SUMMARY:
Preliminary study to compare IntelliVent-ASV to conventional modes used from intubation to extubation or death in ICU patients requiring mechanical ventilation measuring duration of mechanical ventilation in order to design a multicenter large trial.

ELIGIBILITY:
Inclusion criteria:

- Unselected ICU patients invasively ventilated for less than 24 hours, with an expected duration of MV longer than 48 hours.

Exclusion criteria:

* broncho-pleural fistula
* dyshemoglobulinémia
* moribund patient
* do-not-resuscitate order
* chronic respiratory failure requiring long term ventilation,
* patient ventilated more than 24 hours before admission,
* pregnancy,
* age below 18 years,
* protected patients,
* patient already participating in the study,
* Cheynes-Stockes breathing.
* Included patients with a treatment withdrawal decision within 24 hours after inclusion will be excluded,
* patients transferred to another ICU,
* patients needing ECMO, patients randomized to IntelliVent having less than 20% of time in IntelliVent-ASV.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-12; Primary Completion 2013-12 (Actual); Study Completion 2015-01-30 (Actual)

PRIMARY OUTCOMES:
Numbers of manual adjustments | participants are followed until they no longer need ventilation, up to 10 days
  Numbers of manual adjustments of the FULLY CLOSED-LOOP VENTILATION device ( INTELLIVENT ASV)

SECONDARY OUTCOMES:
sedation duration, | participants are followed until they no longer need ventilation, up to 10 days
ventilation parameters | participants are followed until they no longer need ventilation, up to 10 days
Sedation doses | participants are followed until they no longer need ventilation, up to 10 days
Duration of invasive ventilation | participants are followed until they no longer need ventilation, up to 10 days
ICU Mortality | participants are followed until they no longer need ventilation, up to 10 days
28 days mortality | participants are followed until they no longer need ventilation, up to 10 days

CONTACTS AND LOCATIONS:
Locations (2):
- Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer, Toulon, Paca, France
- Anestesia e Rianimazione 2, Fondazione IRCCS Policlinico S. Matteo, Pavia, Lombardy, Italy